CLINICAL TRIAL: NCT02986425
Title: OPERAM: OPtimising thERapy to Prevent Avoidable Hospital Admissions in the Multimorbid Older People: a Cluster Randomised Controlled Trial
Brief Title: OPtimising thERapy to Prevent Avoidable Hospital Admissions in the Multimorbid Older People
Acronym: OPERAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Cork University Hospital (Other); UMC Utrecht (Other); University of Basel (Other); Université Catholique de Louvain (Other); Utrecht University (Other); University of Bern (Other); European Commission (Other); State Secretariat for Education Research and Innovation, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1181-9400
Record Dates: First submitted 2016-10-21; First posted 2016-12-08 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: 3 or More Chronic Conditions for 6 Months or Longer; 5 or More Regular Drugs
Keywords: Drug Utilization Review; Older people
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STRIP intervention (Experimental): The intervention will take place during the initial hospital admission (Index Hospitalisation) or an equivalent situation for outpatients. STRIP is a structured method to perform pharmacotherapy optimisation. The STRIP-intervention consists of 9 steps.
  Interventions: Other: STRIP intervention
- Control (Sham Comparator): Participants in the control group will receive medication review by the prescribing physicians in accordance with usual care. If an extended drug review is in place in a ward/specialty corresponding characteristics are collected on cluster level.
  Interventions: Other: Control

INTERVENTIONS:
Other: STRIP intervention — The STRIP intervention consists of 9 steps:
  1. structured history taking of medication
  2. recording medication and diagnoses in STRIPA
  3. structured drug review based on the STRIPA with the integrated Screening Tool of Older Person's Prescriptions (STOPP)/ Screening Tool to Alert Doctors to the Right Treatment (START) criteria
  4. communication and discussion of the structured drug review with prescribing physician with possible adaptation of the recommendation
  5. shared decision-making with the patient with possible adaptation of the recommendation
  6. optional revision based on new accumulating data during hospitalisation (e.g. new diagnoses, adverse drug reactions)
  7. generation of general practioner (GP) report
  8. delivery of the report to the patient and to the GP (optional additional direct communication)
  9. follow-up
  Other Names: Systematic drug review
  Arms: STRIP intervention
Other: Control — Standard care in the department where the trial is conducted. To keep the patients and the blinded team members blinded one questionnaire will be conducted by the intervention team in both arms. This is considered a SHAM intervention.
  Other Names: Standard care
  Arms: Control

SUMMARY:
The objective of this Randomised Controlled Trial (RCT) is to evaluate whether the Systematic Tool to Reduce Inappropriate Prescribing (STRIP) including STRIP assistant (STRIPA) implemented by an appropriately qualified team will lead to an improvement in clinical and economic outcomes among patients aged 70 years and more with multimorbidity and polypharmacy.

DETAILED DESCRIPTION:
Background:

Drug-related morbidity and mortality is an increasing problem in European healthcare systems. Multimorbidity, polypharmacy and old age are important risk factors for drug-related hospital admissions (DRA). The reported incidence of DRAs in the elderly may be as high as 30% of all acute cases, and about half of DRAs are likely to be preventable. They are mainly related to prescribing problems and non-compliance with drug regimens. A significant proportion of healthcare costs are spent on unnecessary interventions and inappropriate medications. The Systematic Tool to Reduce Inappropriate Prescribing (STRIP) is a structured method to perform a medication review to optimise pharmacotherapy.

Design:

European multi-centre, cluster randomised, controlled trial of people aged 70 years or older, with multimorbidity and polypharmacy, being on an ambulatory visit or on a hospital stay in one of the four participating centres in Ireland, Belgium, Switzerland and the Netherlands. A cluster is defined around a treating physician, i.e. the treating physician is randomised and defines the allocation of his patients. Clusters of patients will be randomised to the intervention arm receiving STRIP for optimising therapy or to the control arm undergoing usual clinical care. The patients of physicians who are allocated to the intervention group will undergo a systematic drug review and pharmacotherapy optimisation by a physician and a pharmacist using STRIP, including the STRIPA software. That provides the research team with a recommendation of changes in the patient's medication. Based on STRIPA recommendation and agreement on changes to the patients' pharmacotherapy between the team of the research physician and pharmacist and the prescribing physician, will the patient receive structured counselling about his/her medication; general practitioners will receive a report. Patients will be further followed for 1 year with follow-up phone calls after 2, 6 and 12 months. For the purpose of this trial, all hospitalisations during follow-up of participants will be adjudicated to assess their relationship to adverse drug events.

Objectives:

The primary objective is to assess the effect of a structured medication review and pharmacotherapy optimisation using the STRIP on drug-related hospitalisations (DRA) caused by over-, mis-, and underuse or over-, mis-, and underprescribing of medications.

Secondary objectives will be to assess the impact of pharmacotherapy optimisation on falls, quality of life, polypharmacy, medication changes, activities of daily living, and mortality.

Statistical considerations:

80 clusters with a cluster size ranging from 12 to 38 participants will be included. Therefore, 2000 patients, 1000 patients in each arm, will be recruited over 18 months. The trial will have 80% power with this sample size.

The primary analysis will be an intention-to-treat (ITT) analysis, whereby all randomised patients will be included in the group they were allocated to.

The primary outcome of drug-related admission will be analysed using a random-effects competing risk proportional hazards model that accounts for the competing risk of death and for clustering of data within centre and prescribing physician.

Overall survival will be analysed using a random-effects Cox proportional hazards model that accounts for clustering of data within centre and prescribing physician. The analysis of falls will also take into account the competing risk of death. Continuous outcomes will be analysed by random-effects linear regression. All effect measures will be accompanied by 95% confidence intervals and all p-values will be two-sided.

ELIGIBILITY:
Inclusion Criteria:

* People 70 years of age or older
* Multimorbidity: 3 or more coexistent chronic conditions defined by 3 distinct International Classification of Diseases (ICD-10) codes with an estimated duration of 6 months or more or based on a clinical decision
* Polypharmacy i.e. five or more different regular drugs (defined as authorised medications with registration numbers) for more than 30 days.
* In inpatient: Estimated minimal length of stay within the cluster is sufficient to apply the intervention
* If outpatient: prescribing physician has GP function and has a planned appointment to conduct intervention

Exclusion Criteria:

* Inability to provide informed consent or to obtain informed consent from a proxy for patients with cognitive impairment
* Direct admission to palliative care (< 24h after admission)
* Has passed or will pass a systematic structured drug review during this hospitalisation or within the last two months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2009 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Patients with confirmed DRA after discharge from the index hospitalisation | 12 months
  The primary outcome is defined as the first confirmed DRA after discharge from the index hospitalisation within a period of 12 months.
  Confirmation of a drug-related hospital admission will be assessed by an independent and blinded adjudication committee (per site). Prolongation of the index hospitalisation and prolongation of any following hospitalisations will not be adjudicated for drug-relatedness. Adjudication is done according to specific guidelines.

SECONDARY OUTCOMES:
Number of survivors | 12 months
  Including causes of death
Number of cancer deaths | 12 months
  As subgroup of all deaths this is considered a negative control outcome.
Number of patients with hospitalisations | 12 months
  Detected during the follow-up phone calls
Number of patients with falls | 12 months
  Detected during the follow-up phone calls
Patients' degree of poly-pharmacy | 12 months
  Degree of polypharmacy, defined as the number of regular long-term medications
Patients' quality of life | 12 months
  Quality of life as measured by the visual analogue scale of the European Quality of Life-5 Dimensions instrument (EQ-5D)
Patients' level of pain/discomfort | 12 months
  Item form EQ-5D questionnaire
Patients' basic activities of daily living | 12 months
  Measured by questionnaire Barthel Index Basic Activities of Daily Living (ADL)
Patients' drug compliance | 12 months
  Measured by the Morisky Medication Adherence Questionnaire (MMAS-8)
Number of clinically significant drug-drug interactions | 2 months
  Assessed based on using STRIPA including the list of diagnosis form the Index Hospitalisation and the updated medication list at follow-up. Assessment will be done at the end of the trial, when all data was collected
Number of drug overuse | 2 months
  Assessed based on using STRIPA including the list of diagnosis form the Index Hospitalisation and the updated medication list at follow-up. Assessment will be done at the end of the trial, when all data was collected
Number of drug underuse | 2 months
  Assessed based on using STRIPA including the list of diagnosis form the Index Hospitalisation and the updated medication list at follow-up. Assessment will be done at the end of the trial, when all data was collected
Number of potentially inappropriate medications | 2 months
  Assessed based on using STRIPA including the list of diagnosis form the Index Hospitalisation and the updated medication list at follow-up. Assessment will be done at the end of the trial, when all data was collected
Number of patients with a serious adverse event | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, Prof., Principal Investigator — Head of Ambulatory Care Department of General Internal Medicine Inselspital, Bern University Hospital, University of Bern, Switzerland; and Institute of Primary Health Care (BIHAM), University of Bern
Locations (4):
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Dept. of Medicine (Geriatrics), University College Cork, Cork, Ireland
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- University of Bern and University Hospital Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data will be deposited in the Bern Open Repository and Information System (BORIS) (www.boris.unibe.ch). BORIS allows searching and is indexed by search engines. All items are stored with a unique Digital Object Identifier (DOI) that can be referenced in respective publication.
  The whole study database in csv format, and will include README files, metadata, information about the performed processing and analytical steps, variable definitions, and references to vocabularies used to help secondary users to understand and reuse the data.
  Data will only be shared upon request. Data use proposals will be evaluated by the OPERAM publication committee.
  The data is owned by the sponsor-investigators. In case of data sharing, a data sharing agreement between the external party and the sponsor-investigator will need to be agreed on and signed.

REFERENCES:
- [Background] Leendertse AJ, Egberts AC, Stoker LJ, van den Bemt PM; HARM Study Group. Frequency of and risk factors for preventable medication-related hospital admissions in the Netherlands. Arch Intern Med. 2008 Sep 22;168(17):1890-6. doi: 10.1001/archinternmed.2008.3. PMID 18809816
- [Background] Gillespie U, Alassaad A, Henrohn D, Garmo H, Hammarlund-Udenaes M, Toss H, Kettis-Lindblad A, Melhus H, Morlin C. A comprehensive pharmacist intervention to reduce morbidity in patients 80 years or older: a randomized controlled trial. Arch Intern Med. 2009 May 11;169(9):894-900. doi: 10.1001/archinternmed.2009.71. PMID 19433702
- [Background] Howard RL, Avery AJ, Slavenburg S, Royal S, Pipe G, Lucassen P, Pirmohamed M. Which drugs cause preventable admissions to hospital? A systematic review. Br J Clin Pharmacol. 2007 Feb;63(2):136-47. doi: 10.1111/j.1365-2125.2006.02698.x. Epub 2006 Jun 26. PMID 16803468
- [Background] Laws MB. Adverse drug reactions as cause of admission to hospital: definition of adverse drug reactions needs to include overdose. BMJ. 2004 Aug 21;329(7463):459-60; author reply 460. doi: 10.1136/bmj.329.7463.459-b. No abstract available. PMID 15321917
- [Derived] Stuber MJ, Brockhus LA, Spinewine A, O'Mahony D, Jennings E, Dalleur O, Knol W, Koek HL, Baggio S, Rodondi N, Aubert CE. Central Nervous System-Active Medications and Risk of Hospital Readmission in Older Multimorbid Adults. J Am Geriatr Soc. 2025 Oct;73(10):3113-3122. doi: 10.1111/jgs.70049. Epub 2025 Aug 29. PMID 40879205
- [Derived] Moutzouri E, Beglinger S, Feller M, Eichenberger A, Dalleur O, Knol W, Emmelot-Vonk M, O'Mahony D, Boland B, Aubert CE, Chocano-Bedoya PO, Aujesky D, Spinewine A, Rodondi N. Inappropriate vitamin D supplementation among multimorbid older patients: a multicountry analysis. BMC Geriatr. 2025 Jul 19;25(1):541. doi: 10.1186/s12877-025-06189-w. PMID 40684074
- [Derived] Gastens V, Chiolero A, Feller M, Bauer DC, Rodondi N, Del Giovane C. Development and internal validation of a new life expectancy estimator for multimorbid older adults. Diagn Progn Res. 2025 Mar 4;9(1):5. doi: 10.1186/s41512-025-00185-9. PMID 40033449
- [Derived] Sibille FX, de Saint-Hubert M, Henrard S, Aubert CE, Goto NA, Jennings E, Dalleur O, Rodondi N, Knol W, O'Mahony D, Schwenkglenks M, Spinewine A. Benzodiazepine Receptor Agonists Use and Cessation Among Multimorbid Older Adults with Polypharmacy: Secondary Analysis from the OPERAM Trial. Drugs Aging. 2023 Jun;40(6):551-561. doi: 10.1007/s40266-023-01029-1. Epub 2023 May 23. PMID 37221407
- [Derived] Sallevelt BTGM, Egberts TCG, Huibers CJA, Ietswaart J, Drenth-van Maanen AC, Jennings E, O'Mahony C, Jungo KT, Feller M, Rodondi N, Sibille FX, Spinewine A, van Puijenbroek EP, Wilting I, Knol W. Detectability of Medication Errors With a STOPP/START-Based Medication Review in Older People Prior to a Potentially Preventable Drug-Related Hospital Admission. Drug Saf. 2022 Dec;45(12):1501-1516. doi: 10.1007/s40264-022-01237-5. Epub 2022 Nov 1. PMID 36319944
- [Derived] Huibers CJA, Sallevelt BTGM, Heij JMJO, O'Mahony D, Rodondi N, Dalleur O, van Marum RJ, Egberts ACG, Wilting I, Knol W. Hospital physicians' and older patients' agreement with individualised STOPP/START-based medication optimisation recommendations in a clinical trial setting. Eur Geriatr Med. 2022 Jun;13(3):541-552. doi: 10.1007/s41999-022-00633-5. Epub 2022 Mar 15. PMID 35291025
- [Derived] Sallevelt BTGM, Huibers CJA, Heij JMJO, Egberts TCG, van Puijenbroek EP, Shen Z, Spruit MR, Jungo KT, Rodondi N, Dalleur O, Spinewine A, Jennings E, O'Mahony D, Wilting I, Knol W. Frequency and Acceptance of Clinical Decision Support System-Generated STOPP/START Signals for Hospitalised Older Patients with Polypharmacy and Multimorbidity. Drugs Aging. 2022 Jan;39(1):59-73. doi: 10.1007/s40266-021-00904-z. Epub 2021 Dec 8. PMID 34877629
- [Derived] Blum MR, Sallevelt BTGM, Spinewine A, O'Mahony D, Moutzouri E, Feller M, Baumgartner C, Roumet M, Jungo KT, Schwab N, Bretagne L, Beglinger S, Aubert CE, Wilting I, Thevelin S, Murphy K, Huibers CJA, Drenth-van Maanen AC, Boland B, Crowley E, Eichenberger A, Meulendijk M, Jennings E, Adam L, Roos MJ, Gleeson L, Shen Z, Marien S, Meinders AJ, Baretella O, Netzer S, de Montmollin M, Fournier A, Mouzon A, O'Mahony C, Aujesky D, Mavridis D, Byrne S, Jansen PAF, Schwenkglenks M, Spruit M, Dalleur O, Knol W, Trelle S, Rodondi N. Optimizing Therapy to Prevent Avoidable Hospital Admissions in Multimorbid Older Adults (OPERAM): cluster randomised controlled trial. BMJ. 2021 Jul 13;374:n1585. doi: 10.1136/bmj.n1585. PMID 34257088
- [Derived] Kempen TGH, Bertilsson M, Hadziosmanovic N, Lindner KJ, Melhus H, Nielsen EI, Sulku J, Gillespie U. Effects of Hospital-Based Comprehensive Medication Reviews Including Postdischarge Follow-up on Older Patients' Use of Health Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e216303. doi: 10.1001/jamanetworkopen.2021.6303. PMID 33929523
- [Derived] Crowley EK, Sallevelt BTGM, Huibers CJA, Murphy KD, Spruit M, Shen Z, Boland B, Spinewine A, Dalleur O, Moutzouri E, Lowe A, Feller M, Schwab N, Adam L, Wilting I, Knol W, Rodondi N, Byrne S, O'Mahony D. Intervention protocol: OPtimising thERapy to prevent avoidable hospital Admission in the Multi-morbid elderly (OPERAM): a structured medication review with support of a computerised decision support system. BMC Health Serv Res. 2020 Mar 17;20(1):220. doi: 10.1186/s12913-020-5056-3. PMID 32183810
- [Derived] Adam L, Moutzouri E, Baumgartner C, Loewe AL, Feller M, M'Rabet-Bensalah K, Schwab N, Hossmann S, Schneider C, Jegerlehner S, Floriani C, Limacher A, Jungo KT, Huibers CJA, Streit S, Schwenkglenks M, Spruit M, Van Dorland A, Donze J, Kearney PM, Juni P, Aujesky D, Jansen P, Boland B, Dalleur O, Byrne S, Knol W, Spinewine A, O'Mahony D, Trelle S, Rodondi N. Rationale and design of OPtimising thERapy to prevent Avoidable hospital admissions in Multimorbid older people (OPERAM): a cluster randomised controlled trial. BMJ Open. 2019 Jun 3;9(6):e026769. doi: 10.1136/bmjopen-2018-026769. PMID 31164366